CLINICAL TRIAL: NCT00746447
Title: Double-blind, Double-dummy, Randomised, Multicentre, 12-months, Comparative Study of the Efficacy and Tolerability of Once Daily 3.0 g Mesalazine Granules vs. Once Daily 1.5 g Mesalazine Granules vs. Three Times Daily 0.5 g Mesalazine Granules for Maintenance of Remission in Patients With Ulcerative Colitis
Brief Title: Once Daily (OD) Versus Three Times Daily (TID) Dosing With Mesalazine Granules for Prevention of Recurrence of Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAG-27/UCR; EudraCT No.: 2004-001218-15
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Colitis, Ulcerative; Recurrence
Keywords: maintenance; 5-ASA; mesalamine; mesalazine; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Recurrence | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3.0g OD (Experimental)
  Interventions: Drug: mesalamine granules
- 1.5g OD (Experimental)
  Interventions: Drug: mesalamine granules
- 0.5g TID (Active Comparator)
  Interventions: Drug: mesalamine granules

INTERVENTIONS:
Drug: mesalamine granules — 3.0g mesalamine in the morning, 0.5g placebo at lunch, 0.5g placebo in the evening;
  Other Names: Salofalk granules; Mesalazine
  Arms: 3.0g OD
Drug: mesalamine granules — 1.5g mesalamine and 1.5g placebo in the morning, 0.5g placebo at lunch, 0.5g placebo in the evening;
  Other Names: Salofalk granules; Mesalazine
  Arms: 1.5g OD
Drug: mesalamine granules — 0.5g mesalamine and 2.5g placebo in the morning, 0.5g mesalamine at lunch, 0.5g mesalamine in the evening
  Other Names: Salofalk granules; Mesalazine
  Arms: 0.5g TID

SUMMARY:
This study intends to study the efficacy and tolerability of once daily 3.0 g mesalazine granules vs. once daily 1.5 g mesalazine granules vs. three times daily 0.5 g mesalazine granules for maintenance of remission in patients with ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Men or women aged 18 to 75 years,
* Historically confirmed diagnosis of ulcerative colitis by endoscopy and histology,
* Patient being in remission, defined (according to Rachmilewitz) as:

Clinical Activity Index (CAI) <= 4, and Endoscopic Index (EI) < 4,

* Extent of inflammation during last acute episode was >15 cm beyond the anal margin,
* Last acute episode ended within 3 months prior to study entry.

Exclusion Criteria:

* Crohn's disease,
* Prior bowel resection leading to diarrhoea,
* Toxic megacolon,
* Gastric or duodenal ulcer,
* Haemorrhagic diathesis,
* Presence of symptomatic organic disease of the gastrointestinal tract (with the exception of haemorrhoids or hiatal hernia),
* Active colorectal cancer or a history of colorectal cancer,
* Serious other secondary illnesses of an acute or chronic nature,
* Asthma,
* Severe impairment of renal (e.g., serum creatinine > 1.5 mg/dl) and/or liver functions (e.g., serum transaminase [ALT and/or AST] or alkaline phosphatase >=2x upper limit of normal [ULN]),
* Application of immunosuppressants within 3 months and/or corticosteroids (oral, intravenous [IV] or topical rectal) within 30 days prior to baseline,
* Application of non-steroidal anti-inflammatory drugs (NSAIDs) as long term treatment (i.e. > 6 weeks), other than acetylsalicylic acid (<= 350 mg/day), or paracetamol,
* Known intolerance/hypersensitivity to salicylic acid and its derivatives or to any of the other constituents of the study drugs,
* Well-founded doubt about the patient's cooperation,
* Existing or intended pregnancy, breast-feeding,
* Women of child-bearing potential without adequate contraceptive protection, e.g., hormonal contraception, intrauterine device (IUD), double-barrier method of contraception (e.g., use of a condom and spermicide), partner has undergone vasectomy and subject is in monogamous relationship. The investigator is responsible for determining whether the subject has adequate birth control for study participation,
* Participation in another clinical trial within the last 30 days,simultaneous participation in another clinical trial, or previous participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients still in clinical remission at the final/withdrawal examination, with clinical relapse defined as a CAI >4 with an increase of ≥3 points from baseline. | week 52 or premature withdrawal

SECONDARY OUTCOMES:
Time to relapse | within 52 weeks
Proportion of patients in endoscopical remission, defined as a mucosal appearance score of ≤ 1 at final/withdrawal examination. | week 52 or premature withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mueller, Dr., Study Director — Dr. Falk Pharma GmbH
Locations (1):
- Evangelisches Krankenhaus Kalk, Medical Dept., Cologne, Germany

REFERENCES:
- [Result] Kruis W, Jonaitis L, Pokrotnieks J, Mikhailova TL, Horynski M, Batovsky M, Lozynsky YS, Zakharash Y, Racz I, Kull K, Vcev A, Faszczyk M, Dilger K, Greinwald R, Mueller R; International Salofalk OD Study Group. Randomised clinical trial: a comparative dose-finding study of three arms of dual release mesalazine for maintaining remission in ulcerative colitis. Aliment Pharmacol Ther. 2011 Feb;33(3):313-22. doi: 10.1111/j.1365-2036.2010.04537.x. Epub 2010 Dec 8. PMID 21138455